CLINICAL TRIAL: NCT07102420
Title: Understanding Artificial Intelligence Anxiety Within Different Physical Activity Profiles: Comparing Athletes and Sedentary Individuals
Brief Title: Artificial Intelligence Anxiety Within Different Physical Activity Profiles
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/053
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-07

CONDITIONS: Athletes; Sedanter
Keywords: physical activity; artificial intelligence anxiety; athletes
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sedentary individuals: Sedentary individuals who have not engaged in regular exercise within the past six months, who have been exposed to basic concepts of artificial intelligence (through media, news, education, etc.), who possess sufficient cognitive ability to complete the questionnaires, and who do not have any chronic neurological, orthopedic, cardiovascular, or psychological conditions.
  Interventions: Other: Questionnaire and Physical Exam
- Athletes: Licensed athletes who have engaged in regular exercise or sports at least twice a week during the past six months, who have been exposed to basic concepts of artificial intelligence (through media, news, education, etc.), who possess sufficient cognitive capacity to complete the questionnaires, and who do not have any chronic neurological, orthopedic, cardiovascular, or psychological conditions.
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Artificial Intelligence Anxiety Scale

SUMMARY:
The aim of this study is to compare artificial intelligence anxiety (AIA) in athletes and sedentary individuals, evaluate its relationship with exercise frequency, and identify the subdimensions that cause high anxiety at the level of AIA scale items.

DETAILED DESCRIPTION:
The study will include healthy individuals aged between 18 and 45 years who either engage in regular exercise or lead a sedentary lifestyle. Participants with regular exercise or sports habits and those who are sedentary will be compared in terms of their anxiety levels toward artificial intelligence. Prior to assessment, written informed consent will be obtained from all participants. Additionally, demographic and health-related data will be collected, including age, sex, weight, height, presence of chronic diseases, medication use, history of surgical operations, frequency of daily activities, pain status, and alcohol or tobacco use. Data collection will be conducted using the Artificial Intelligence Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 45 years of age
* Having engaged in regular exercise or sports at least twice a week over the past six months (for athlete group)
* Not having engaged in regular exercise during the past six months (for sedentary group)
* Being exposed to basic concepts of artificial intelligence (via media, news, education, etc.)
* Having sufficient cognitive ability to complete the questionnaires

Exclusion Criteria:

* Having a chronic neurological, orthopedic, cardiovascular, psychological, or similar medical condition
* Having a serious physical disability that prevents participation in exercise
* Incomplete or inconsistent responses in the questionnaires
* Having undergone a recent surgical operation
* Lack of voluntary consent to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study plans to include healthy individuals aged 18 to 45 years, consisting of both regularly exercising participants and sedentary individuals.
Sampling Method: Non-Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Artificial Intelligence Anxiety Scale | baseline
  The Artificial Intelligence Anxiety Scale (AIAS) is an assessment tool that asks each participant to reflect on their current experiences. It is a 7-point Likert-type scale, ranging from 1 (not at all) to 7 (completely). The scale consists of four subdimensions: learning, job replacement, socio-technical blindness, and AI configuration. The total score ranges from a minimum of 21 to a maximum of 147. Higher scores indicate higher levels of anxiety experienced in relation to artificial intelligence.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Akkoyun Sert, PhD, Study Chair — KTO Karatay University; Fatma Çiftçi, PhD, Study Chair — KTO Karatay University
Locations (1):
- Kto Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No